CLINICAL TRIAL: NCT05822180
Title: Evaluation of the Efficacy and Safety of Nano-S1 in Adult Patients Infected With SARS-Cov-2: "COVID Nano-S1
Brief Title: Evaluation of the Efficacy and Safety of Nano-S1
Acronym: COVNANOS1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: General Administration of Military Health, Tunisia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COVID NANO S1
Record Dates: First submitted 2023-04-19; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2022-01

CONDITIONS: COVID-19 Pneumonia
Keywords: ARGENT COLLOIDAL

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A bras actif (Experimental): The experimental arm has received the Nanos product orally with a dose of 30mL, 3 times per day and away from meals (2 hours after a meal or on an empty stomach).
  Interventions: Drug: NANOS1 , argent colloïdal ,
- B bras controle (Placebo Comparator): The placebo arm has received the Nanos product orally with a dose of 30mL, 3 times per day and away from meals (2 hours after a meal or on an empty stomach).
  Interventions: Drug: NANOS1 , argent colloïdal ,

INTERVENTIONS:
Drug: NANOS1 , argent colloïdal , — orally, during 5 day

SUMMARY:
This study aims to assess the efficacy of the efficacy and safety of investigational drug (NanoS) in patients with mild to moderate COVID-19 at high risk for progression to severe COVID-19, including death.

DETAILED DESCRIPTION:
We conducted a prospective randomized double-blind clinical trial over five months to determine the efficacy of NanoS compared to placebo. The effectiveness of treatment was measured by the significant decline in the number of cases of covid-19 infection and/or a decrease in the viral load determined by SARS-CoV-2 cycle threshold (Ct) value using RT-PCRs test.

ELIGIBILITY:
Inclusion Criteria:

1. Participants are hospitalized in a COVID unity or outpatient follow-up by the investigator
2. Participants who have positive SARS-CoV-2 test result and the onset of symptoms of COVID-19 ≤7 days prior to randomization, Not exceed the 7th day since the beginning of disease symptoms; and the randomization's day.
3. Present at least one of these symptoms: Participants who have one or more mild or moderate COVID-19 symptoms: Fever, general signs such as: headaches, asthenia, myalgia, arthralgia, etc... ENT signs such as: Sore throat, anosmia, agueusia, hypoacusis, deafness, etc... Digestive signs such as: diarrhea, vomiting, abdominal pain, etc... Respiratory signs such as: dyspnea, cough, etc... And cutaneous signs such as: skin rash, livedo, etc...
4. Present an oxygen saturation patients with SpO2 > 94% at room air
5. Present at least one of these risk factors:

   Participants who satisfy one or more than one of the following high risks for progression to severe COVID-19, including death: Age 65 years old Or -Age between 18 and 64 years old with at least one of these risk factors: Obesity (BMI> 30 kg/m2),and/or diabetes under treatment and/or cardiovascular disease (including hypertension and stable angina) high blood pressure

   and/or Chronic obstructive pulmonary disease (COPD) disease and/or asthma and/or Neoplasia (solid tumour; hematological malignancy) neoplasia, and/or a blood disease and/or heart failure and/or chronic renal failure (Cl creat> 30Mml/min) and/or unstabe angina and/or autoimmune disease.
6. Have signed the informed consent to participate in this trial.

Exclusion Criteria:

* Non observance.Non-compliant patient With drawal of Consent. Patient who refuses blood samples.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
Clinical evolution | 14DAY
  The evolution clinical state of evaluated patient clinical state after 14 days since the beginning of the disease is made with " a 8-point ordinal scale " (WHO Rd Blue print novel Coronavirus
  / COVID-19 Therapeutic Trial Synopsis / 18 February 2020)

SECONDARY OUTCOMES:
Disappearance of clinical signs | 3 days
  Disappearance of clinical signs (functional and physical) reported and confirmed at the study inclusion visit (Visit 1). The deadline of disappearance:
  - Less than or equal to 3 days
Viral load Ct value | admission ,DAY6, DAY14
  Evaluate the significative decrease of viral load between DAY 0 and DAY 6, and between DAY6 and DAY14 by the variation of CtT values.
Negativation of the RT- PCR | DAY 14
  Negativation of the RT- PCR after 14 days since the beginning of the disease. of the randomization
Tolerance | DAY 14, DAY 30
  Évaluate the tolerance of the study product (Nano-S1) versus placebo on the occurrence of adverse events
Systemic passage | DAY 30
  6. Evaluate the systemic passage of the product of the study by the assay in the blood on J1 (before taking PI ID), on J6 (on the last day) and on DAY 30 in the two study groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Agili Faida, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No